CLINICAL TRIAL: NCT06084143
Title: Analysis of Suicide Dynamics in Link to the COVID-19 Pandemic
Acronym: DSL-Covid-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9026
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
Keywords: Covid-19; Suicide
MeSH Terms: conditions — COVID-19; Suicide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Covid is a virus that first appeared in China in 2019 and was quickly described as a pandemic virus by its globalized nature. The unprecedented occurrence of the virus has led to several health and restrictive government measures. The Covid-19 pandemic and health measures have been able to contribute to the deterioration of the mental health of citizens as it has already been observed during the former pandemic context (Sars covid in 2003 in China or the Spanish flu).

Among the consequences of a negative impact on mental health, investigators assume that there is an increase in transitions to the completed suicidal act. However, current studies and observations tend to note that there has been no major change in the dynamics of successful suicides during the Covid period.

However, there are biases in the studies conducted: some suicide deaths may have been hidden and not reported as such, due to several factors. For example, the measure of the evolution of suicide attempts that was most often made by the measure of the evolution of the number of hospitalizations for this reason can be a source ofestimate whether people who did this gesture were not hospitalized after a visit to the emergency room or if they gave up attending because of the pandemic. Moreover, suicide deaths are more difficult to report as such when they occur at home than after hospitalization.

It is therefore interesting to study the dynamics of suicide during this health crisis retrospectively based on data from the Strasbourg Institute of Forensic Medicine containing the census of the Alsace region, which was hit hard by the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Died between 01/01/2018 and 12/31/2021
* Absence of opposition from the patient expressed in writing during his lifetime to the reuse of his personal data for scientific research purposes.

Exclusion Criteria:

* Presence of opposition by the patient expressed in writing during his lifetime to the reuse of his personal data for scientific research purposes.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient died between 01/01/2018 and 12/31/2021
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-07-21 (Estimated); Study Completion 2024-07-21 (Estimated)

PRIMARY OUTCOMES:
Suicide rates before and after the Covid-19 pandemic | from January 1, 2018 to December 31, 2021

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Psychiatrie - CHU de Strasbourg - France, Strasbourg, France